CLINICAL TRIAL: NCT05347303
Title: Effects of Finding-oriented Orthopedic Manual Therapy Combined With Foam Roller on Lower Limb Flexibility and Muscular Power in Colombian University Athletes: a Randomized Controlled Clinical Trial
Brief Title: Orthopedic Manual Therapy vs Foam Roller on Flexibility, Joint Range of Motion, rm and Vertical Jump
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: "University of Jaén"
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Athletes
Keywords: Orthopedic Manual Therapy; Foam roller; Strength

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Epidat randomization will be used to assign the groups. This assignment will be hidden, so the therapists will not be aware of which group each subject belongs to. Random assignment will be done by an investigator who will have no influence on the measurements or statistical analysis. The analysis will be carried out by another researcher who will remain unrelated to the measurements and the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group (EG) after taking initial measurements and signing their informed consent will be subjected to an 8-week intervention plan with 2 sessions per week where they will receive 1 MTOH and 1 Foam roller on discontinuous days. MTOH consists of first evaluating the structures that have restrictions, whether soft tissues or joints, to later be treated with a specific manual technique. For this, evaluation methods based on Kaltenborn are used when it comes to joints and Pilat when focusing on soft tissues. Interventions will not exceed 20 minutes per subject. For the foam roller, subjects will perform slides on the instrument using their body weight on the following muscles: quadriceps, hamstrings, gastrocnemius, and tensor fascia lata, for 60 seconds with 3 repetitions for each. Each repetition will have a rest period of 30 seconds, this will be done on both lower limbs.
  Interventions: Other: Finding-oriented orthopedic manual therapy treatment combined with foam roller
- Control group (Active Comparator): After taking measurements, they will perform 2 foam roller sessions per week following the same indications expressed in the experimental group.
  Interventions: Other: Foam roller treatment

INTERVENTIONS:
Other: Finding-oriented orthopedic manual therapy treatment combined with foam roller — Blind randomized controlled clinical trial, where a total of 87 people, men and women, of legal age, university athletes of collective disciplines will be evaluated. The experimental group will receive foam roller therapy and manual therapy guided by findings (n = 44) for 8 weeks.
  Arms: Experimental group
Other: Foam roller treatment — Subjects will perform slides on the instrument using their body weight on the following muscles: quadriceps, hamstrings, gastrocnemius, and tensor fascia lata, for 60 seconds with 3 repetitions for each. Each repetition will have a rest period of 30 seconds, this will be done on both lower limbs.
  Arms: Control group

SUMMARY:
Orthopedic Manual Therapy (OMT) is one of the branches of physiotherapy that has less evidence about its action and efficacy, but those who have had the opportunity to apply or receive it know its great benefits. Currently, worldwide, the approach given to physiotherapy goes hand in hand with the guidelines of the TMO, but in Colombia it is not seen in the same way. The objective of this TFM is to compare the effects of Finding-Oriented Orthopedic Manual Therapy combined with Foam Roller versus the effects of Foam Roller alone, specifically in terms of muscle power and lower limb flexibility in Colombian athletes. For this, a randomized controlled clinical trial will be carried out with two groups that will undergo different interventions. To measure the variables, the CMJ jump protocol will be used with the Optogait and the Wells or sit and reach test.

DETAILED DESCRIPTION:
This research corresponds to an experimental study, a blind randomized controlled clinical trial, where a total of 87 people, men and women, of legal age, university athletes of collective disciplines, distributed in 2 groups will be evaluated: the experimental group will receive therapy with foam roller and with manual therapy guided by findings-oriented (n = 44) for 8 weeks, while the control (n = 43) will only receive the foam roller treatment. The variables will be measured with equipment and protocols validated in both groups. Evaluations will be made at the beginning of the intervention and immediately after the end of this period, all the data being unified in an Excel, assigning a code to each individual to maintain the privacy of the participants. As independent variables, sociodemographic data will be taken, as a result variable, the Maximum Repetition (RM) will be obtained following the protocol of a maximum repetition, the range of joint mobility using the goniometer pro app on an iPhone XR, flexibility with the Sit & Reach in V and the vertical jump measured with OptoGait. All variables will be measured pre and post intervention. As a result, manual therapy is expected to generate greater effects on the sports performance of university athletes in collective disciplines. Based on statistical processes, the data will be processed and it will be evaluated whether or not there are significant differences within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Be active in any of the joint sports programs of the Fundación Universitaria del Área Andina headquarters Pereira - Colombia.
* Voluntarily accept participation in the study.
* Sign the consent informed.

Exclusion Criteria:

* Have a lower limb injury that may affect flexibility or muscle power.
* Refuse to participate in the study.
* Be under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-17 (Actual)

PRIMARY OUTCOMES:
Flexibility | Up to twelve weeks
  The sit and reach or Wells test is a test commonly used to measure the flexibility of the hamstring muscles and the posterior muscles in general (Mayorga-Vega et al., 2014). This test will be carried out following the guidelines of the American College of Sports Medicine (American College of Sport Medicine [ACSM], 2000). This test consists of placing the person evaluated sitting on the floor in front of a box with their feet resting on it without any type of footwear, keeping their knees fully extended, on the box there is a plate with a tape measure on which the person evaluated must place their hands, later they will perform a maximum trunk flexion trying to cover the greatest possible distance with their upper limbs without altering the rest of the position, if the person cannot reach the plate, the missing distance will be measured to be able to contact it and it will be presented as a negative value.
Joint range of motion | Up to twelve weeks
  The goniometer pro application available for iphone will be used. This tool has been previously tested and validated in the Latino population (Barboza et al., 2020). For this, the mobile device will be located with a system of straps that will ensure the position of the equipment on the segment to generate the displacement, once the individual is located in the starting position, the initial point will be selected in the application to then carry out the movement. The mobile device will then measure the displacement and give a measurement in degrees (°) that will be recorded.
Muscular Power | Up to twelve weeks
  The Optogate will be used, following the CMJ jump test, in which the subject stands in the middle of the instrument's optical led strips, adopts a position of knee and hip flexion where the knee joint forms an angle of 90 °, to ensure that it will be done in this way, it will be measured with a manual goniometer and a rope will be placed to give the subject a stimulus when he is in the correct position. In addition, you must place your hands on the waist and execute the jump in a single movement, fluid and without interruptions, before taking the measurements the subject will be allowed to become familiar with the test, in the first session. On measurement days, 3 jumps will be allowed and the one with the highest score will be considered valid.
Muscle strength | Up to twelve weeks
  Strength will be measured through the 1RM test, validated in different populations, regardless of gender or age (Grgic, Lazinica, Schoenfeld, & Pedisic, 2020). For the calculation of 1RM, the subjects will first receive an adaptation session, where they will get used to the gesture with low load so that after 2 days they can perform the real test. The actual test will consist of a warm-up with low resistance performing 10 repetitions of the exercise, then the load will be progressively increased until failure occurs, regardless of the verbal reinforcement given. A repetition will be considered successful when the subject performs the full range of motion without significant fasciculations or compensatory movements. The RM will be determined in 5 attempts for all subjects, all following the guidelines of the National Strength and Conditioning Association (Baechele & Earle, 2008).

CONTACTS AND LOCATIONS:
Locations (1):
- Andina Area University Foundation, Pereira, Colombia

REFERENCES:
- [Derived] Afanador-Restrepo DF, Rodriguez-Lopez C, Rivas-Campo Y, Baena-Marin M, Castellote-Caballero Y, Quesada-Ortiz R, Osuna-Perez MC, Carcelen-Fraile MDC, Aibar-Almazan A. Effects of Myofascial Release Using Finding-Oriented Manual Therapy Combined with Foam Roller on Physical Performance in University Athletes. A Randomized Controlled Study. Int J Environ Res Public Health. 2023 Jan 12;20(2):1364. doi: 10.3390/ijerph20021364. PMID 36674120